CLINICAL TRIAL: NCT01163565
Title: A Prospective Randomized Equivalence Trial to Evaluate the Safety of the Ligasure in Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Todd McMullen, Associate Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00004394
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Multinodular Goitre; Grave's Disease; Thyroid Nodule
Keywords: Thyroidectomy
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ligasure device (Active Comparator)
  Interventions: Device: Ligasure Device
- Hand ties (No Intervention)

INTERVENTIONS:
Device: Ligasure Device — Ligasure device used to seal blood vessels during left or right side of a total thyroidectomy. Traditional method of hand ties/clips on contralateral side.
  Arms: Ligasure device

SUMMARY:
This is a randomized, prospective equivalence trial on the safety of the Ligasure Vessel Sealing System as used in thyroid surgery. The Ligasure system is a hand held surgical device that uses heat to seal blood vessels during surgery. It has been a tested and accepted technology in abdominal surgery and it is now being applied to surgery of the thyroid gland because it is faster than the traditional method of tying blood vessels that a surgeon must do manually. To remove the thyroid gland safely the surgeon must dissect the gland away from the recurrent laryngeal nerve which controls the vocal cords and patient's voice. Protecting this nerve is the key step in all thyroid surgery as its damage can permanently alter a patient's voice and even obstruct the airway. At this time the worldwide accepted rate of nerve injury is 2 in 100 patients. The hypothesis of this study is that the nerve injury rates for surgery using the Ligasure device are similar to that seen when surgeons manually tie blood vessels. The investigators protocol will evaluate the function of the recurrent laryngeal nerve after removing the thyroid gland using the Ligasure device in comparison to the traditional method where the surgeon manually ties blood vessels. In this study, for patients undergoing total thyroidectomy for a benign condition, each patient will be randomized to have one lobe of thyroid (left or right) removed using manual tying of blood vessels and the other side will have the surgeon use the Ligasure device to seal blood vessels. Every patient has a pre- and post-operative independent assessment of vocal cord function using nasopharyngoscopy to ensure that the vocal cords are working normally prior to surgery and also to document vocal cord dysfunction if there is an injury to the recurrent laryngeal nerve. The investigators intent is to show that the Ligasure system is a safe method to sealing vessels in thyroid surgery and that the thermal dispersion of this device does not pose a significant increase in risk to the recurrent laryngeal nerve

DETAILED DESCRIPTION:
Diathermy is an accepted modality to aid surgery and maintain hemostasis and is used in all forms of surgery including head and neck, neurosurgery and general surgery. The Ligasure vessel sealing system uses heat energy and has been approved for use in many different types of surgery and has been tested and accepted for use in multiple countries, including Canada. What is being tested in this proposal is the application of this accepted technology to thyroid surgery. There has been one previous randomized trial examining the Ligasure device in thyroid surgery but this was designed to look at operative times and bleeding episodes in comparison to manually tying blood vessels. It has been proven that the Ligasure device makes operations quicker and is just as effective at sealing blood vessels as manual tying by the surgeon. However, in thyroid surgery injury to the recurrent laryngeal nerve is an important concern as the nerve is in close proximity to the gland. Damage to the nerve could temporarily or permanently alter a patient's voice making it hoarse. In this study we examine if the heat generated by the device could damage the recurrent laryngeal nerve if it is held close enough for prolonged time periods. There are case reports that indicate that the Ligasure is safe but this study intends in a prospective, randomized manner to prove that the use of the Ligasure system does not affect nerve injury rates compared to a surgeon manually tying blood vessels during thyroid surgery.

Our hypothesis is that the use of the Ligasure vessel sealing system in thyroid surgery is as safe as the traditional manual tying of blood vessels by the surgeon in terms of injury to the recurrent laryngeal nerve.

We propose a randomized, prospective equivalence trail to compare recurrent laryngeal nerve injury rates with the use of the Ligasure device or manually tying blood vessels. The thyroid gland has two lobes, a left and a right, and under each lobe there is the recurrent laryngeal nerve (thus two per patient). With the traditional manual tying of vessels, approximately 2% of patients will have altered function in one of the recurrent laryngeal nerve, and we expect that the rates of altered function in the Ligasure patient cohort to be the same. To prove this we will enroll patients with benign thyroid disease, including multinodular goitre, Grave's disease, thyroid nodule or thyroiditis, having total thyroidectomy. Excluded are patients under 18 and those with known cancer as well as those undergoing reoperative surgery or those with known recurrent laryngeal nerve dysfunction. The patients will be randomized by computer to have dissection of the thyroid gland on one side (left or right) done with the traditional manual tying method and the other side will be done with the surgeon using the hand-held Ligasure device. The randomization process uses a random number generator to assign the patient a number as they are booked for the operating theatre. This process is independent of the surgeon such that they do not know the side to use the Ligasure until the day of the operation. After surgery an independent assessment of the vocal cords with nasopharyngoscopy is done on both the left and right side within 6 weeks of surgery by an otolaryngologist that is blinded to the surgical technique. This allows us to determine if either the left or right recurrent laryngeal nerve has been injured. If there is an injury it will be linked to whether the surgeon manually tied the vessels on that side or if they used the Ligasure device. Sample size calculations for this equivalence trial were based on Blackwelder (Controlled Clinical Trials 1982;3:345-353) which outline that to detect a 5% difference in injury rates, set at 2 in 100, between the Ligasure and traditional techniques we will need to complete dissections on 96 patients (each patient has one side Ligasure and one side manual tying).

ELIGIBILITY:
Inclusion Criteria:

* multinodular goiter
* Grave's disease
* thyroid nodule

Exclusion Criteria:

* thyroid carcinoma
* reoperative surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-04; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
recurrent laryngeal nerve injury | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Walter C Mackenzie Health Sciences Centre, Edmonton, Alberta, Canada